CLINICAL TRIAL: NCT02548377
Title: Remote Ischemic Preconditioning in Head and Neck Cancer Reconstruction - A Randomized Controlled Trial
Acronym: RIPC-HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Andreas Engel Krag, M.D., Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPC-HNC
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms; Surgical Flaps; Ischemic Preconditioning; Hemostasis; Thrombosis; Immune System; Reperfusion Injury
MeSH Terms: conditions — Head and Neck Neoplasms; Thrombosis; Reperfusion Injury | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Experimental): Four 5-minute cycles of upper extremity ischemia, each separated by five minutes of reperfusion. The treatment will be carried out with a tourniquet inflated to 200 mmHg during general anaesthesia prior to flap ischemia and transfer.
  Interventions: Procedure: Remote ischemic preconditioning
- Sham (Sham Comparator): The tourniquet will be attached to the patient's upper extremity but never inflated.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Remote ischemic preconditioning
  Arms: Remote ischemic preconditioning
Procedure: Sham
  Arms: Sham

SUMMARY:
The purpose of the trial is to investigate, if remote ischemic preconditioning reduces the risk of complications in patients undergoing resection of head and neck cancer and immediate reconstruction with autologous free tissue transfer.

Remote ischemic preconditioning is a treatment, which is carried out by inducing brief episodes of upper arm occlusion using an inflatable tourniquet.

Blood samples will be taken during the operation and postoperatively to evaluate the effects of remote ischemic preconditioning. These blood samples will be analyzed for clotting properties and markers of inflammation.

Furthermore, effects on the blood supply of the transferred tissue flap will be measured by infrared thermography.

Effects on surgical complication rates will be obtained by clinical follow-up and patient chart review.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified or clinically suspected malignant tumor in the oral cavity, maxillae, mandible, pharynx, larynx, and/or esophagus.
* Will undergo tumor resection and immediate free flap reconstruction at Aarhus University Hospital, Denmark.
* The reconstruction is planned with a single free flap.

Exclusion Criteria:

* Arterial and/or venous thromboembolism within the last three months.
* The reconstruction is planned with more than one free flap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Acute effects on primary hemostasis: Reduced collagen-induced platelet aggregation in whole blood measured by the Multiplate Analyzer. | Blood samples will be analyzed immediately. Data will be assessed and presented within five years.

SECONDARY OUTCOMES:
Acute effects on secondary hemostasis: Plasma samples will be analyzed by standard coagulation assays. | Plasma samples will be analyzed immediately. Data will be assessed and presented within five years.
Acute effects on fibrinolysis: Plasma samples will be analyzed for markers of fibrinolysis. | Data will be analyzed, assessed, and presented within five years.
Acute effects on global hemostasis: Plasma samples will be analyzed with the thrombin generation assay. | Data will be analyzed, assessed, and presented within five years.
Acute effects on systemic inflammation: Plasma samples will be analyzed for complement, acute-phase proteins, cytokines, and leukocytes. | Data will be analyzed, assessed, and presented within five years.
Effects on complication rates: Flap complications, systemic complications, morbidity and mortality. | Follow-up is 30 days from the operation. Data will be obtained from visits to the outpatient clinic and by patient chart review. Data will be analyzed, assessed, and presented within five years.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, M.D., Ph.D., Study Chair — Aarhus University Hospital
Locations (1):
- Centre for Hemophilia and Thrombosis, Department of Clinical Biochemistry, Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Background] Taylor GI, Palmer JH. The vascular territories (angiosomes) of the body: experimental study and clinical applications. Br J Plast Surg. 1987 Mar;40(2):113-41. doi: 10.1016/0007-1226(87)90185-8. PMID 3567445
- [Background] Chubb DP, Taylor GI, Ashton MW. True and 'choke' anastomoses between perforator angiosomes: part II. dynamic thermographic identification. Plast Reconstr Surg. 2013 Dec;132(6):1457-1464. doi: 10.1097/01.prs.0000434407.73390.82. PMID 24281576
- [Background] Selber JC, Angel Soto-Miranda M, Liu J, Robb G. The survival curve: factors impacting the outcome of free flap take-backs. Plast Reconstr Surg. 2012 Jul;130(1):105-113. doi: 10.1097/PRS.0b013e318254b1b9. PMID 22418714
- [Background] Khouri RK, Cooley BC, Kunselman AR, Landis JR, Yeramian P, Ingram D, Natarajan N, Benes CO, Wallemark C. A prospective study of microvascular free-flap surgery and outcome. Plast Reconstr Surg. 1998 Sep;102(3):711-21. doi: 10.1097/00006534-199809030-00015. PMID 9727436
- [Background] Culliford AT 4th, Spector J, Blank A, Karp NS, Kasabian A, Levine JP. The fate of lower extremities with failed free flaps: a single institution's experience over 25 years. Ann Plast Surg. 2007 Jul;59(1):18-21; discussion 21-2. doi: 10.1097/01.sap.0000262740.34106.1b. PMID 17589253
- [Background] Olsson E, Svartling N, Asko-Seljavaara S, Lassila R. Activation of coagulation and fibrinolysis during reconstructive microsurgery in patients with cancer. Microsurgery. 2001;21(5):208-13. doi: 10.1002/micr.1040. PMID 11494394
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Background] Schmidt MR, Smerup M, Konstantinov IE, Shimizu M, Li J, Cheung M, White PA, Kristiansen SB, Sorensen K, Dzavik V, Redington AN, Kharbanda RK. Intermittent peripheral tissue ischemia during coronary ischemia reduces myocardial infarction through a KATP-dependent mechanism: first demonstration of remote ischemic perconditioning. Am J Physiol Heart Circ Physiol. 2007 Apr;292(4):H1883-90. doi: 10.1152/ajpheart.00617.2006. Epub 2006 Dec 15. PMID 17172279
- [Background] Kerendi F, Kin H, Halkos ME, Jiang R, Zatta AJ, Zhao ZQ, Guyton RA, Vinten-Johansen J. Remote postconditioning. Brief renal ischemia and reperfusion applied before coronary artery reperfusion reduces myocardial infarct size via endogenous activation of adenosine receptors. Basic Res Cardiol. 2005 Sep;100(5):404-12. doi: 10.1007/s00395-005-0539-2. Epub 2005 Jun 17. PMID 15965583
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849
- [Background] Dickson EW, Reinhardt CP, Renzi FP, Becker RC, Porcaro WA, Heard SO. Ischemic preconditioning may be transferable via whole blood transfusion: preliminary evidence. J Thromb Thrombolysis. 1999 Aug;8(2):123-9. doi: 10.1023/a:1008911101951. PMID 10436142
- [Background] Lim SY, Yellon DM, Hausenloy DJ. The neural and humoral pathways in remote limb ischemic preconditioning. Basic Res Cardiol. 2010 Sep;105(5):651-5. doi: 10.1007/s00395-010-0099-y. Epub 2010 May 7. PMID 20449597
- [Background] Addison PD, Neligan PC, Ashrafpour H, Khan A, Zhong A, Moses M, Forrest CR, Pang CY. Noninvasive remote ischemic preconditioning for global protection of skeletal muscle against infarction. Am J Physiol Heart Circ Physiol. 2003 Oct;285(4):H1435-43. doi: 10.1152/ajpheart.00106.2003. Epub 2003 Jun 5. PMID 12791590
- [Background] Ropcke DM, Hjortdal VE, Toft GE, Jensen MO, Kristensen SD. Remote ischemic preconditioning reduces thrombus formation in the rat. J Thromb Haemost. 2012 Nov;10(11):2405-6. doi: 10.1111/j.1538-7836.2012.04914.x. No abstract available. PMID 22947090
- [Background] Pedersen CM, Cruden NL, Schmidt MR, Lau C, Botker HE, Kharbanda RK, Newby DE. Remote ischemic preconditioning prevents systemic platelet activation associated with ischemia-reperfusion injury in humans. J Thromb Haemost. 2011 Feb;9(2):404-7. doi: 10.1111/j.1538-7836.2010.04142.x. No abstract available. PMID 21083644
- [Background] Mounsey RA, Pang CY, Boyd JB, Forrest C. Augmentation of skeletal muscle survival in the latissimus dorsi porcine model using acute ischemic preconditioning. J Otolaryngol. 1992 Oct;21(5):315-20. PMID 1469751
- [Background] Kuntscher MV, Schirmbeck EU, Menke H, Klar E, Gebhard MM, Germann G. Ischemic preconditioning by brief extremity ischemia before flap ischemia in a rat model. Plast Reconstr Surg. 2002 Jun;109(7):2398-404. doi: 10.1097/00006534-200206000-00034. PMID 12045567
- [Background] Kuntscher MV, Kastell T, Sauerbier M, Nobiling R, Gebhard MM, Germann G. Acute remote ischemic preconditioning on a rat cremasteric muscle flap model. Microsurgery. 2002;22(6):221-6. doi: 10.1002/micr.10041. PMID 12375286
- [Background] Moses MA, Addison PD, Neligan PC, Ashrafpour H, Huang N, Zair M, Rassuli A, Forrest CR, Grover GJ, Pang CY. Mitochondrial KATP channels in hindlimb remote ischemic preconditioning of skeletal muscle against infarction. Am J Physiol Heart Circ Physiol. 2005 Feb;288(2):H559-67. doi: 10.1152/ajpheart.00845.2004. Epub 2004 Sep 30. PMID 15458954
- [Background] Restifo RJ, Thomson JG. The preconditioned TRAM flap: preliminary clinical experience. Ann Plast Surg. 1998 Oct;41(4):343-7. doi: 10.1097/00000637-199810000-00001. PMID 9788213
- [Background] Kraemer R, Lorenzen J, Kabbani M, Herold C, Busche M, Vogt PM, Knobloch K. Acute effects of remote ischemic preconditioning on cutaneous microcirculation--a controlled prospective cohort study. BMC Surg. 2011 Nov 23;11:32. doi: 10.1186/1471-2482-11-32. PMID 22111972
- [Background] Kolbenschlag J, Sogorski A, Harati K, Daigeler A, Wiebalck A, Lehnhardt M, Kapalschinski N, Goertz O. Upper extremity ischemia is superior to lower extremity ischemia for remote ischemic conditioning of antero-lateral thigh cutaneous blood flow. Microsurgery. 2015 Mar;35(3):211-7. doi: 10.1002/micr.22336. Epub 2014 Oct 3. PMID 25278482